CLINICAL TRIAL: NCT00087113
Title: A Phase II Evaluation Of Pemetrexed (ALIMTA, LY231517, IND #40061) In the Treatment Of Recurrent Carcinoma Of The Cervix
Brief Title: Pemetrexed Disodium in Treating Patients With Recurrent Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0127T; LILLY-H3E-US-JMGS
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Cancer
Keywords: cervical squamous cell carcinoma; recurrent cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Pemetrexed

INTERVENTIONS:
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well pemetrexed disodium works in treating patients with recurrent cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of pemetrexed disodium in patients with recurrent carcinoma of the cervix that failed higher priority treatment protocols.
* Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Beginning 7 days before and continuing until 3 weeks after the last dose of pemetrexed disodium, patients also receive oral folic acid daily and cyanocobalamin (vitamin B_12) intramuscularly every 9 weeks.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 22-60 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the cervix

  * Squamous cell or non-squamous cell
  * Recurrent disease
  * Progressive disease
* Measurable disease

  * At least 1 unidimensionally measurable target lesion ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR ≥ 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are considered non-target lesions unless disease progression is documented or a biopsy is obtained to confirm persistence at least 90 days after completion of radiotherapy
* Not amenable to surgery, radiotherapy, or other therapy
* Must have received 1 prior systemic chemotherapy regimen for persistent or recurrent squamous cell or non-squamous cell carcinoma of the cervix

  * Chemotherapy administered with primary radiotherapy as a radiosensitizer is not considered a systemic chemotherapy regimen
* Not eligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* AST and ALT ≤ 3 times upper limit of normal (ULN)*
* Alkaline phosphatase ≤ 3 times ULN*
* Bilirubin ≤ 1.5 times ULN NOTE: * ≤ 5 times ULN if liver metastases are present

Renal

* Creatinine clearance ≥ 45 mL/min

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* Neuropathy (sensory and motor) ≤ grade 1
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic or immunologic agents for the malignant tumor
* At least 24 hours since prior growth factors
* One prior non-cytotoxic (biologic or cytostatic) regimen for recurrent or persistent disease allowed, including, but not limited to, the following:

  * Monoclonal antibodies
  * Cytokines
  * Small-molecule inhibitors of signal transduction
* No concurrent routine colony-stimulating factors

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No more than 1 prior cytotoxic chemotherapy regimen with either single or combination cytotoxic drug therapy
* No prior pemetrexed disodium

Endocrine therapy

* At least 1 week since prior hormonal therapy for the malignant tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered
* No prior radiotherapy to > 25% of bone marrow

Surgery

* Recovered from prior surgery

Other

* At least 3 weeks since other prior therapy for the malignant tumor
* No nonsteroidal anti-inflammatory drugs for 2-5 days before, during, and for 1-2 days after study drug administration

  * Concurrent daily low-dose (≤ 325 mg/day) aspirin therapy allowed
* No prior therapy that would contraindicate study participation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Antitumor activity
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (22):
- United States (22):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Doctors Medical Center, Modesto, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Women's Cancer Center - Las Vegas, Las Vegas, Nevada
  - SUNY Downstate Medical Center, Brooklyn, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Williamette Gynecologic Oncology P.C., Salem, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Miller DS, Blessing JA, Bodurka DC, Bonebrake AJ, Schorge JO; Gynecologic Oncology Group. Evaluation of pemetrexed (Alimta, LY231514) as second line chemotherapy in persistent or recurrent carcinoma of the cervix: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2008 Jul;110(1):65-70. doi: 10.1016/j.ygyno.2008.03.009. Epub 2008 May 5. PMID 18455781